CLINICAL TRIAL: NCT01010763
Title: A Prospective Controlled Multi-Center Study on M2a Magnum Total Hip Arthroplasty
Brief Title: A Study on M2a Magnum Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT.CR.RROW2
Record Dates: First submitted 2009-11-05; First posted 2009-11-10 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Degenerative Joint Disease; Avascular Necrosis
MeSH Terms: conditions — Joint Diseases; Osteonecrosis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- M2a Magnum (Experimental): Total HIp Arthroplasty using with the M2a Magnum Large Metal Articulation is an ultra-high performance metal-on-metal articulation with a big ball (greater than or equal to 38mm) in acetabulums as small as 44mm.
  Interventions: Device: Total Hip Arthroplasty
- M2a Taper (Active Comparator): Total Hip Arthroplasty using with the M2a Taper Acetabular System consists of a titanium outer shell with cobalt chromium (Co-Cr-Mo) metallic liner, which articulates with with a cobalt chromium (Co-Cr-Mo) modular femoral head.
  Interventions: Device: Total Hip Arthroplasty

INTERVENTIONS:
Device: Total Hip Arthroplasty — Degenerated hip is replaced with implantable devices, which include femoral stem, acetabular cup, femoral head and acetabular liner(control group only).

SUMMARY:
The purpose of this study includes the investigation of Metal-ion release and Renal Function analysis in M2a Total Hip Arthroplasty.

DETAILED DESCRIPTION:
There are no clinical studies conducted on its performance in Asian population. Furthermore clinical data is required to support marketing and validate design of M2A Magnum.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for primary Total Hip Replacement
* Patients aged over 20
* Patients with limited co-morbidity- ASA I-III
* Patients must be able to understand instructions and be willing to return for follow-up
* Patients willing to provide blood and urine samples for metal ion analysis at follow-up

Exclusion Criteria:

* Pre-existing metal implants
* Infection, sepsis, and osteomyelitis
* Uncooperative patient or pt with neurologic disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* osteomalacia
* distant foci of infections which may spread to the implant site
* rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* vascular insufficiency, muscular atrophy, or neuromuscular disease
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Ozono, M.D., Ph.D., Principal Investigator — Kansai Rosai Hospital
Locations (1):
- Kansai Rosai Hospital, Amagasaki, Hyogo Pref., Japan

REFERENCES:
- [Derived] Ando W, Yamamoto K, Atsumi T, Tamaoki S, Oinuma K, Shiratsuchi H, Tokunaga H, Inaba Y, Kobayashi N, Aihara M, Ohzono K. Comparison between component designs with different femoral head size in metal-on-metal total hip arthroplasty; multicenter randomized prospective study. J Orthop. 2015 Jun 10;12(4):228-36. doi: 10.1016/j.jor.2015.05.008. eCollection 2015 Dec. PMID 26566324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Period of Recruitment was from December 2009 until December 2011. Recruitements were done at medical clinics by providing detailed explanation of procedure as well as study protocol, including randomization & right of withdrawal.
Pre-assignment Details: Four patients withdrer before randomization.
Period: Overall Study
Arm/Group | M2a Magnum | M2a Taper
Started | 96 | 84
Completed | 61 | 54
Not Completed | 35 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | M2a Magnum | M2a Taper | Total
Number analyzed (Participants) | 96 | 84 | 180
Age, Continuous [Mean (Full Range); unit: years] | 65 [39 to 86] | 67 [41 to 98] | 66 [39 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 61 | 133
  Male | 24 | 23 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 96 | 84 | 180
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 96 | 84 | 180
Harris Hip Score [Mean (Full Range); unit: units on a scale] — Harris Hip Score is physician assessing hip functional scoring system, which includes 4 components (pain, function, deformity and range of motion) with minimum score of 0 & maximum score of 100.
  Maximum & Minimum score of each subscale is pain: 0-44, function: 0-47, Deformity: 0-4 and Range of motion: 0-5.
  Current report uses summed score of each patient to compare total Harris Hip Score.
  Higher score means better outcomes. Population: Preoperative Harris Hip Score of two patients in Magnum arm were failed to obtain.
  units on a scale
    number analyzed (Participants) | 94 | 84 | 178
    (all) | 52.3 [3 to 79] | 51.2 [22 to 82] | 51.7 [3 to 82]
EQ-5D [Mean (Full Range); unit: units on a scale] — EQ-5D is patient reported outcome measure to score patient's health related quality of life with minimum score of -0.111 and maximum score of 1.000.
  Higher score means better outcomes. Population: Preoperative EQ-5D questionnaire was not completed by two subjects (one subject each arm).
  units on a scale
    number analyzed (Participants) | 95 | 83 | 178
    (all) | 0.620 [-0.109 to 1.000] | 0.647 [0.049 to 1.000] | 0.633 [-0.109 to 1.000]
UCLA Activity Score [Mean (Full Range); unit: units on a scale] — UCLA is physician assessing scoring system to assess patient's activity level. Minimum score is 0 (completely inactive) and maximum score is 9 (Regularly participates in impact sports) with 1 point increments depending on patient's activity level.
  Higher score means higher activity level achieved.
  units on a scale | 3.1 [1 to 6] | 3.0 [2 to 6] | 3.0 [1 to 6]

OUTCOME MEASURES:

1. Primary Outcome: Range of Motion
Description: Hip Flexion Angle at 1 year postoperatively
Time Frame: 1 year
Population: 2 patients in M2a Magnum group and 4 patients in M2a Taper group were failed to obtain Range of Motion data at 1 year follow-up visit.
Measure: Mean (Full Range); unit: degrees
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 94 | 80
degrees | 109.2 [70 to 130] | 110.2 [70 to 130]

2. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 3 month
Population: 3 patients in M2a Taper group were failed to obtain Metal Ion data at 3 month follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 96 | 81
microgram/Litter | 0.7 [0 to 2.3] | 0.9 [0 to 2.7]

3. Secondary Outcome: UCLA Activity Score
Description: UCLA is physician assessing scoring system to assess patient's activity level. Minimum score is 0 (completely inactive) and maximum score is 9 (Regularly participates in impact sports) with 1 point increments depending on patient's activity level.
  Higher score means higher activity level achieved.
Time Frame: 5 year
Population: 59 patients in M2a Magnum group and 59 patients in M2a Taper group were failed to obtain UCLA Activity Score data at 5 year follow-up visit.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 37 | 25
units on a scale | 4.97 [3 to 9] | 4.8 [1 to 8]

4. Secondary Outcome: Radiographic Assessment
Description: number of participants, whose x-ray shows any signs of radiographic changes (osteolysis, heterotopic ossification and/or radiolucency)
Time Frame: 5 year
Population: 45 patients in M2a Magnum group and 36 patients in M2a Taper group were failed to be assessed radiographically at 5 year follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 51 | 48
Participants
  Acetabular Osteolysis | 0 | 0
  Acetabular Radiolucency | 0 | 0
  Stem Osteolysis | 0 | 0
  Stem Radiolucency | 2 | 7
  Heterotopic Ossification | 2 | 1
  no abnormalities | 47 | 40

5. Secondary Outcome: Harris Hip Score
Description: Harris Hip Score is physician assessing hip functional scoring system, which includes 4 components (pain, function, deformity and range of motion) with minimum score of 0 & maximum score of 100.
  Maximum & Minimum score of each subscale is pain: 0-44, function: 0-47, Deformity: 0-4 and Range of motion: 0-5.
  Current report uses summed score of each patient to compare total Harris Hip Score.
  Higher score means better outcomes.
Time Frame: 5 year
Population: 68 patients in M2a Magnum group and 62 patients in M2a Taper group were failed to obtain Harris Hip Score data at 5 year follow-up visit.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 28 | 22
units on a scale | 96.3 [72 to 100] | 94.5 [64 to 100]

6. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 6 month
Population: 4 patients in M2a Taper group were failed to obtain Metal Ion data at 6 month follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 96 | 80
microgram/Litter | 0.9 [0 to 5.1] | 1.2 [0 to 8.9]

7. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 1 year
Population: 7 patients in M2a Magnum group and 9 patients in M2a Taper group were failed to obtain Metal Ion data at 1 year follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 89 | 75
microgram/Litter | 1.2 [0 to 12.9] | 1.8 [0 to 15.4]

8. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 2 year
Population: 12 patients in M2a Magnum group and 10 patients in M2a Taper group were failed to obtain Metal Ion data at 2 year follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 84 | 74
microgram/Litter | 1.2 [0.13 to 6.3] | 2.0 [0.2 to 11.0]

9. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 3 year
Population: 21 patients in M2a Magnum group and 19 patients in M2a Taper group were failed to obtain Metal Ion data at 3 year follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 75 | 65
microgram/Litter | 0.98 [0 to 4.9] | 2.9 [0 to 44.0]

10. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 4 year
Population: 50 patients in M2a Magnum group and 46 patients in M2a Taper group were failed to obtain Metal Ion data at 4 year follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 46 | 38
microgram/Litter | 1.09 [0.11 to 4.0] | 3.1 [0 to 22.0]

11. Secondary Outcome: Metal Ion
Description: Blood Cobalt Ion Concentration 0 was imputed for the measurement result being below detection limit.
Time Frame: 5 year
Population: 33 patients in M2a Magnum group and 30 patients in M2a Taper group were failed to obtain Metal Ion data at 5 year follow-up visit.
Measure: Mean (Full Range); unit: microgram/Litter
Arm/Group | M2a Magnum | M2a Taper
Number analyzed (Participants) | 63 | 54
microgram/Litter | 1.07 [0.11 to 7.6] | 3.8 [0.16 to 71.0]

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | M2a Magnum | M2a Taper
All-Cause Mortality (participants affected / at risk) | 0/96 | 3/84
Serious Adverse Events (participants affected / at risk) | 1/96 | 1/84
Other Adverse Events (participants affected / at risk) | 2/96 | 3/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M2a Magnum (N=96) | M2a Taper (N=84)
Revision due to Adverse Reaction to Metal Debris (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femoral Epicondyle Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M2a Magnum (N=96) | M2a Taper (N=84)
Dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Cerebral Infarction (Vascular disorders) | 1 (1) | 0 (0)
Intra-operative fracture (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-21): https://cdn.clinicaltrials.gov/large-docs/63/NCT01010763/Prot_SAP_000.pdf